CLINICAL TRIAL: NCT04355520
Title: A Phase Ib, Single-arm, Open-label Study of TQ-B3525 Tablets Combined With Fulvestrant Injection in Subjects With HR-positive, HER2-negative and PIK3CA Mutation Advanced Breast Cancer
Brief Title: A Study of TQ-B3525 Tablets Combined With Fulvestrant Injection in Subjects With HR-positive, HER2-negative and PIK3CA Mutation Advanced Breast Cancer
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3525-I-02
Record Dates: First submitted 2020-04-20; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-02

CONDITIONS: HR-positive, HER2-negative and PIK3CA Mutation Advanced Breast Cancer
MeSH Terms: interventions — TQ-B3525; Fulvestrant

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3525 tablets combined with fulvestrant injection (Experimental): TQ-B3525 tablets were taken orally, once daily in 28-day cycle; fulvestrant injection 500mg administered intravenously (IV) on day 1, day 15 of first cycle and on day 1 of follow-up treatment cycle. Each cycle is 28 days.
  Interventions: Drug: TQ-B3525; Drug: Fulvestrant injection

INTERVENTIONS:
Drug: TQ-B3525 — TQ-B3525 tablets were taken orally, once daily in 28-day cycle; The doses were 20 mg and 30 mg.
Drug: Fulvestrant injection — Fulvestrant injection 500mg administered intravenously (IV) on day 1, day 15 of first cycle and on day 1 of follow-up treatment cycle. Each cycle is 28 days.

SUMMARY:
This is a open-label, multicenter phase Ib study to evaluate safety and efficacy of TQ-B3525 tablets combined with fulvestrant injection in subjects with HR-positive, HER2-negative and PIK3CA mutation advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1. Histopathologically confirmed breast cancer. 2. Hormone receptor(HR) positive and human epidermal growth factor receptor-2 (HER2) negative for primary or metastatic tumors confirmed by immunohistochemistry test.

  3. Agree to provide at least 10 unstained sections of tumor tissue obtained within 2 years (surgery or biopsy) for genetic mutation detection and with PIK3CA mutation positive.

  4. Age ≥18 years, postmenopausal women. 5. Inoperable, locally advanced recurrent and/or metastatic tumor, and has at least one measurable lesion.

  6. Inappropriate to receive radical resection or radiation therapy. 7. Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1.

  8. Life expectancy ≥12 weeks. 9. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study.

  10. Understood and signed an informed consent form.

Exclusion Criteria:

* 1. Has known untreated or active CNS metastasis. 2.Previous or co-existing cancers of a different site or histology from primary breast cancer.

  3. Inadequate bone marrow hematopoiesis. 4. Abnormal liver function. 5. Renal abnormalities. 6. Has bleeding risk. 7. Gastrointestinal disorder. 8. Cardio-cerebrovascular anomaly. 9. Previous treatment: A) Has received fulvestrant injection; B) Has received PI3K, AKT and mTOR inhibitors; C) Has received anti-tumor treatment, including chemotherapy, radiotherapy, hormone therapy, biotherapy, immunotherapy, and surgical treatment, less than 4 weeks after the first administration; D) Has received oral targeted drugs less than 5 half-lives to the first administration; E) Has received palliative radiotherapy for non-target lesions within 2 weeks before the first administration; F) Toxicity related to previous anti-tumor treatment did not recover to ≤ grade 1, except for hair loss.

  10.Has participated in other clinical trials within 30 days. 11.Has received major surgical treatment within 1 month or unhealed traumatic injury.

  12. Has a history of organ transplantation or hematopoietic stem cell transplantation within 60 days prior to the first administration.

  13.Immunosuppressant or systemic or absorbable local hormone therapy is required to achieve the aim of immunosuppression (dose > 10mg/ day prednisone or other therapeutic hormones) and is still used within 2 weeks after the first administration.

  14.Active bacterial or fungal infections diseases. 15.Human immunodeficiency virus (HIV) infection. 16.Pregnant or lactating female patients. 17.Has mental and neurological diseases. 18. With severe or poorly controlled diseases. 19. Has a history of active tuberculosis. 20. Patients have inadequate compliance to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2020-07 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) | up to 28 days
  Subjects appear the toxic reaction relate to the drug after treatment within 28 days.

SECONDARY OUTCOMES:
Overall response rate (ORR) assessed by investigator | up to 72 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR).
Disease control rate（DCR） | up to 72 weeks
  Percentage of participants achieving Complete Response (CR) and Partial Response (PR) and Stable Disease (SD).
Duration of Response (DOR) | up to 72 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression based on radiographic assessment.
Progression-free survival (PFS) | up to 72 weeks
  PFS defined as the time from first dose to the first documented progressive disease (PD) or death from any cause.
Overall survival (OS) | up to 72 weeks
  OS defined as the time from the first dose to death from any cause. Participants who do not die at the end of the extended follow-up period, or were lost to follow-up during the study, were censored at the last date they were known to be alive.
Cmax | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on day 1; Hour 0 of day 15; and hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on day 28.
  Cmax is the maximum plasma concentration of TQ-B3525 or metabolite(s).
Tmax | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on day 1; Hour 0 of day 15; and hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on day 28.
  To characterize the pharmacokinetics of TQ-B3525 by assessment of time to reach maximum plasma concentration.
AUC0-t | Hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on day 1; Hour 0 of day 15; and hour 0, 0.5, 1, 2, 3, 4, 6, 8, 11, 24 hours post-dose on day 28.
  To characterize the pharmacokinetics of TQ-B3525 by assessment of time to reach maximum plasma concentration.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Cancer Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Hospital of Jilin university, Changchun, Jilin
  - Liaoning Cancer Hospital, Shenyang, Liaoning